CLINICAL TRIAL: NCT06184061
Title: An Assessment of the Acute Effects of Herbal Dietary Supplements on Aerobic Performance in Recreational Athletes
Brief Title: Acute Effects of Herbal Dietary Supplements on Aerobic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Nezire İnce, Asst. Prof., Eastern Mediterranean University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ETK00-2023-0207
Record Dates: First submitted 2023-11-29; First posted 2023-12-28 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Diet, Healthy
Keywords: Athlete Performance; Nutritional Supplement; Recovery
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Placebo will be given to this group (100ml, contain same carbohydrate amount as herbal supplement)
- Interventional Group (Active Comparator): Herbal Supplement will be given to this group (100ml, Herbal Supplement)
  Interventions: Combination Product: Herbal Supplement

INTERVENTIONS:
Combination Product: Herbal Supplement — Herbal supplement will be the mixture of strawberry, black mulberry, blueberry, raspberry, ginseng, ashwagandha, honey, water
  Arms: Interventional Group

SUMMARY:
Positive effects of herbal supplements such as red berries, ginseng, ashwagandha on athletic performance have been reported. The aim of this study was to evaluate the acute effects of a herbal dietary supplement prepared from a mixture of red berries, ginseng and ashwagandha on aerobic performance of recreational athletes.

DETAILED DESCRIPTION:
In the beginning of the study anthropometric measurements (weight (kg), height (cm), BMI, waist circumference (cm), body fat percentage, lean body mass, skeletal muscle mass) will be taken from the participants who accepted to participate in the study.

During the study, participants will be restricted from consuming alcohol, caffeine, red fruit, ginseng and ashwagandha.

First, Yoyo Intermittent Recovery Level 1 performance test (The Yo-Yo test is a maximal aerobic endurance fitness test, involving running between markers placed 20 meters apart, at increasing speeds, until exhaustion) will be done to all participants In this step, participants will not drink anything. Then there will be a 2-week break.

At the end of the 3-week break, the participants will be divided into two groups by block randomization method and one group will receive a herbal nutritional supplement mixture (100 ml 30 minutes before training). The other group will drink a placebo prepared with the same texture and consistency as our main mixture, containing an equal amount of carbohydrates (100 ml 30 minutes before training). Then the same performance test will be repeated. At the end of the test also 1 and 2 minutes after end of the test, the participants' heart rate measurement will be taken with a finger-type pulse oximeter and recorded . At the end of the test, perceived exertion levels will be questioned using the Borg scale.

ELIGIBILITY:
Inclusion Criteria:

* Being a student in the Exercise and Sports sciences department
* Not using any supplement
* Not being in a period that will affect sleep patterns (midterm/finals week, holiday, etc.)
* Doing regular exercise

Exclusion Criteria:

* Having a known food allergy
* Using any supplement
* Being a professional athlete
* Drinking alcohol regularly

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Vo2 Max | Up to 1 week
  Once the test is completed, participants' Vo2 max values will be calculated using the formula "Vo2 max= Distance covered x 0.0084 + 36.4"
Total distance covered in Yo-Yo intermittent recovery test (level 1) | Up to 1 week
  Once the test is completed, total distance covered by participants during the test will be recorded in meters.

SECONDARY OUTCOMES:
Change between end-test heart rate and heart rate 1 minute post Yo-Yo intermittent recovery test (level 1) | 1 minutes
  Volunteers' heart rate was taken immediately after the Yo-Yo intermittent recovery test (level 1) and 1 minute post test. Heart rates were detected by using finger tip pulse oximeter
Change between end-test heart rate and heart rate 2 minutes post Yo-Yo intermittent recovery test (level 1) | 2 minutes
  Volunteers' heart rate was taken immediately after the Yo-Yo intermittent recovery test (level 1) and 2 minute post test. Heart rates were detected by using finger tip pulse oximeter

OTHER OUTCOMES:
BMI | Up to 2 weeks
  BMI will be calculated. For the calculation of BMI; weight (kg), height (m) will be measured and formulated as follow (weight (kg) / (height (m))2
Waist Circumference | Up to 2 weeks
  Waist circumference of the participants will be measured by placing the measuring tape around your middle at a point halfway between the bottom of your ribs and the top of your hips (just above the belly button) and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Nezire Ince, Study Director — Eastern Mediterranean University
Locations (1):
- Nezire, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No